CLINICAL TRIAL: NCT05185726
Title: Treatment for Preschool Age Children Who Stutter: A Randomised, Multicentre, Non-inferiority Parallel Group Pragmatic Trial With Mini-KIDS, the Social Cognitive Behaviour Therapy and the Lidcombe Program With 249 Children
Brief Title: TreatPaCS = Treatment for Preschool Age Children Who Stutter
Acronym: TreatPaCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas More University of Applied Sciences (Other)
Collaborators: Universiteit Antwerpen (Other); University of Liege (Other); Artevelde University of Applied Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-OHC-210048
Record Dates: First submitted 2021-12-08; First posted 2022-01-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Stuttering, Developmental
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Intervention Model Description: A three arm 1:1:1 randomised, multicentre, open-label non-inferiority parallel group pragmatic trial
Who Masked: Outcomes Assessor
Masking Description: Videos of speech will be scores for %SS by assessors who are blinded for the treatment arm in which the child belongs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mini-KIDS (Experimental): Mini-KIDS is a direct treatment based on principles of stuttering modification, with pseudo-stuttering, that is, deliberate stuttering, as one of the main components. The program for 4-6-year old children consists of four stages: Stage 1 = desensitization, Stage 2 = modification, Stage 3 = identification and Stage 4 = generalization. The program for 2-4-year old children does not include stage 3. Speech therapist and parent(s) are the speech model for the child. They add normal dysfluencies to their speech. Later on in treatment and if necessary, children learn to recognise and alter their stuttering moments.
  Interventions: Behavioral: Mini-KIDS
- Social-Cognitive Behaviour Treatment (Experimental): The social cognitive behaviour therapy contains 5 treatment phases: (1) conditioning speaking activities, (2) cognitive training focused on emotions, (3) cognitive training focused on cognitions, (4) emotional training and (5) skill training (Boey, 2010). This treatment is not directed at the speech of the children, but rather at the cognitive and emotional aspects that surround the stuttering.
  Interventions: Behavioral: Social Cognitive Behavioural Therapy
- Lidcombe Program (Active Comparator): The Lidcombe Program (LP) is an operant program that directly provides verbal feedback to the child's stutter-free speech (mainly) and the child's stuttering (occasionally). The program comprises two stages: Stage 1 in which (near) zero levels of stuttering are achieved and Stage 2 in which the achieved (near) zero levels of stuttering are maintained for a long period of time. The LP usually takes between 11 to 23 (60-minute) treatment sessions to achieve the goals of Stage 1, i. e. (near) zero levels of stuttering.
  Interventions: Behavioral: Lidcombe Program

INTERVENTIONS:
Behavioral: Lidcombe Program — The LP consists of Stage 1 and Stage 2. Stage 1 aims at reducing the stuttering of the PCWS to (near) zero levels of stuttering. During stage 1, parents learn to provide verbal contingencies during daily, 10-minute practice sessions with their PCWS.
  During Stage 1, treatment sessions are scheduled weekly. When the child has typical scores of 0 and 1 on the SR-scale with more 0s than 1s per week for three consecutive weeks, and the stuttering is rated as 0 or 1 during the treatment session, the child can proceed to stage 2.
  The maintenance phase starts when the stuttering is reduced to (near) zero stuttering and parents are able to implement the practice sessions when it is necessary (when stuttering relapses). Treatment sessions to monitor if achieved goals are maintained are scheduled with an interval of 2, 2, 4, 4, 8, 8 and 16 weeks.
  Other Names: LP
  Arms: Lidcombe Program
Behavioral: Mini-KIDS — Mini-KIDS for 4-6-year old PCWS consists of four stages: Stage 1 = desensitization, Stage 2 = identification, Stage 3 = modification and Stage 4 = generalization. The program for 2-4-year old child does not include stage 2. SLT and parent(s) are the speech model for the child. They add normal disfluencies and pseudo-stuttering to their speech at first to make sure the child dares to stutter and the child as well as the parent(s) are desensitized for it. Later on in treatment and if necessary, child learn to recognise and alter their stuttering moments. The maintenance phase starts when the child and parent(s) achieved the goals of Stage 4. Usually the stuttering is reduced to (near) zero stuttering. Treatment sessions to monitor if achieved goals are maintained are scheduled with an interval of 2, 2, 4, 4, 8, 8 and 16 weeks.
  Arms: Mini-KIDS
Behavioral: Social Cognitive Behavioural Therapy — A parent training is organised for parents with children who stutters who receive SCBT.
  The parent training exists of 10 one-hour group evening sessions for parents to discuss and offer education topics about what stuttering is, how stuttering looks like, ...
  The program is delivered in 5 phases and each phase takes as long as is necessary for the PCWS (variable): (1) conditioning speaking activities, (2) cognitive training focused on emotions, (3) cognitive training focused on cognitions, (4) emotional training and (5) skill training.
  The maintenance phase starts when the child and parent(s) achieved the goals of the 5 phases. During the maintenance sessions, the SLT asks the parent(s) to report about the child and observes the speech of the child.
  Other Names: SCBT
  Arms: Social-Cognitive Behaviour Treatment

SUMMARY:
Treatment for preschool age children who stutter: a randomised, multicentre, non-inferiority parallel group pragmatic trial with Mini-KIDS, the social cognitive behaviour therapy and the Lidcombe Program with 249 children

DETAILED DESCRIPTION:
Three treatment approaches for preschool age children who stutter are delivered and %Syllables Stuttered at 18 months post-randomisation of the three arms are compared .

Mini-KIDS is a direct treatment based on principles of stuttering modification, with pseudo-stuttering, that is, deliberate stuttering, as one of the main components. The program for 4-6-year old children consists of four stages: Stage 1 = desensitization, Stage 2 = modification, Stage 3 = identification and Stage 4 = generalization. The program for 2-4-year old children does not include stage 3. Speech therapist and parent(s) are the speech model for the child. They add normal dysfluencies to their speech. Later on in treatment and if necessary, children learn to recognise and alter their stuttering moments.

The social cognitive behaviour therapy contains 5 treatment phases: (1) conditioning speaking activities, (2) cognitive training focused on emotions, (3) cognitive training focused on cognitions, (4) emotional training and (5) skill training (Boey, 2010). This treatment is not directed at the speech of the children, but rather at the cognitive and emotional aspects that surround the stuttering.

The Lidcombe Program (LP) is an operant program that directly provides verbal feedback to the child's stutter-free speech (mainly) and the child's stuttering (occasionally). The program comprises two stages: Stage 1 in which (near) zero levels of stuttering are achieved and Stage 2 in which the achieved (near) zero levels of stuttering are maintained for a long period of time. The LP usually takes between 11 to 23 (60-minute) treatment sessions to achieve the goals of Stage 1, i. e. (near) zero levels of stuttering.

ELIGIBILITY:
Inclusion Criteria:

Preschool age children must

* stutter (identified by the Speech-Language Therapist)
* be aged between 2 - 6.5 years
* have normal hearing reported by the parent(s)
* have, if bilingual, a parent who speaks a language that the SLT understands and speaks to allow clear communication
* have at least one parent agreeing to be intensively involved in treatment and knowing that s/he will implement treatment at home
* have at least one parent who is willing and able to videorecord his/her child regularly

Exclusion Criteria:

- have a syndrome such as Down Syndrome.

Ages: 24 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
% of Syllables Stuttered (%SS) | 18 months post-randomisation
  The %SS at 18 months post-randomisation will be determined in two video samples (at home and in the treatment session) and the average will be used. They will be conpared between the 3 programs.

SECONDARY OUTCOMES:
Severity rating of the stuttering | 3-, 6-, 9-, 12-, 18-months and 2- and 5-year post-randomisation
  The severity rating of the stuttering will be averaged over home and treatment session and will be compared between the 3 programs
Speech attitude (Kiddy CAT) scores | 18-months post-randomisation
  Score on the KiddyCAT will be compared between the 3 programs
Score on Quality of life questionnaire | at 18-months, 2- and 5-years post-randomisation
  Score on the EQ-5D-Y-proxy 2 will be compared between the 3 programs
Score on Impact of Stuttering on Parents and Preschooler (ISPP) questionnaire | at 18-months post-randomisation
  Score on the ISPP will be compared between the 3 programs
% of Syllables Stuttered (%SS) | 3-, 6-, 9-, 12-months and 2- and 5-year post-randomisation
  The %SS will be determined in two video samples (at home and in the treatment session) and the average will be used. They will be conpared between the 3 programs.
Treatment duration (number of hours) | Through study completion, on average 9 months
  Treatment duration will be calculated in number of hours
Treatment duration (number of weeks) | Through study completion, on average 9 months
  Treatment duration will be calculated in number of weeks
Treatment duration (number of sessions) | Through study completion, on average 9 months
  Treatment duration will be calculated in number of weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Van Eerdenbrugh, Dr, Principal Investigator — Thomas More
Locations (1):
- Sabine Van Eerdenbrugh, Antwerp, Belgie, Belgium

IPD SHARING:
Plan to Share IPD: No